CLINICAL TRIAL: NCT00302107
Title: A Placebo-Controlled Study of Mirtazapine for PTSD in OIF/OEF Veterans
Brief Title: A Placebo-Controlled Study of Mirtazapine for PTSD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBA-019-05F; NCT00449189 (obsolete NCT alias)
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Anxiety; PTSD
Keywords: Mirtazapine; PTSD; Veterans; antidepressant
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Mirtazapine
  Interventions: Drug: Mirtazapine
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine — Mirtazapine initiated at 15mg qhs and titrated in 15mg increments to a maximum of 45 mg qhs as tolerated.
  Other Names: Remeron
  Arms: Arm 1
Drug: Placebo — Look-a-like placebo tablets under double-blind conditions
  Arms: Arm 2

SUMMARY:
Objective: To study the efficacy and tolerability of mirtazapine (Remeron) in the treatment of PTSD.

Research Design: This is an 8-week randomized, double-blind, placebo-controlled treatment trial of mirtazapine for the treatment of PTSD as defined on the Clinical Assessment of PTSD Scale (CAPS).

Methodology: After signing an informed consent and meeting all inclusion/exclusion criteria, the patient is randomized to either mirtazapine versus placebo for 8-week duration. During the study a pharmacist maintains the randomization log and verifies the order for the placebo or mirtazapine in look-a-like tablets. Patients' symptoms, side effects and compliance are assessed bi-weekly. Based on symptomology and occurrence of side effects, the investigator increases the medication in 15 mg increments, as tolerated, until a maximum therapeutic benefit is achieved, not to exceed 45 mg/day. The dosing is at bedtime. Compliance is assessed by bi-weekly pill count at week 4 and week 8. Patients are given supportive clinical management during the clinic visits. An investigator is available by telephone 24 hrs a day in case of emergency. Patients may be seen more often if needed. Efficacy will be measured by the following assessment scales: Montgomery-Asberg Depression Rating Scale (MADRS), Hamilton Anxiety Scale (Ham-A), Clinical Global Impression Severity of Illness (CGI-s), Clinical Global Impression of Improvement (CGI-I), Global Assessment of Functioning (GAF), CAPS, Treatment Outcome PTSD rating scale (TOP-8), and Davidson Trauma Scale (DTS).

Clinical Significance: Mirtazapine has shown promise in treating PTSD in an open label trial. This study is the next step in proving mirtazapine's efficacy in treatment of PTSD.

DETAILED DESCRIPTION:
Title: A Placebo-Controlled Study of Mirtazapine for PTSD in OIF/OEF Veterans and Veterans from all other Southwest Asia Conditions

Sponsor of the study: VA Merit grant

Research Setting: Subjects will be recruited from the mental health and primary care outpatient clinics and inpatient units. The informed consent process will be conducted in a private setting. Rating scales and laboratory procedures will also be performed in a private setting.

Purpose of the study including hypothesis to be tested: The primary objective is to evaluate the efficacy and tolerability of mirtazapine (Remeron) in the treatment of PTSD. Primary Hypothesis to be tested: Veterans with PTSD will have improvement in their symptomatology after 8 weeks of treatment with mirtazapine compared to those treated with placebo.

Background, including results of relevant research, gaps in the current knowledge. PTSD is a common mental illness, afflicting about 3 percent of persons, or 12 million North Americans. PTSD is a common consequence of disasters, rape, auto accidents, and violent crime, with about half of trauma victims suffering acute symptoms. One fourth of victims of acute PTSD progress to develop chronic PTSD. Presently, there are only two medications indicated for PTSD (sertraline and paroxetine). Long-term effects of untreated PTSD are serious, including depression, alcohol and drug abuse, violence, and suicide. The VA Healthcare System is a natural clinical laboratory for study of PTSD, since 14 - 30 % of Vietnam Combat Veterans continue to suffer consequences of this disorder. Preliminary clinical data from an open studies and one small placebo-controlled study of mirtazapine in the treatment of PTSD suggests that mirtazapine is effective and may have a unique pharmacological profile in treating PTSD.

Potential Benefits to the research subject and knowledge to be gained: The actual patient participant may benefit from further reduction in underlying psychiatric symptoms. There is substantial potential for knowledge about PTSD treatment to be gained by the cumulative data gathered in this study that may improve the health care of veterans and nonveterans in the future.

Definition of the population to be studied and justification: The population to be studied is outpatient veterans with current PTSD, diagnosed by the use of the MINI. Patients may be recruited from mental health, inpatient units or Primary Care Outpatient Clinics, however; the majority of the study is intended to be outpatient. The justification for use of a PTSD population is that new treatments for PTSD are needed, particularly with combination of medications since monotherapy rarely is fully effective.

Number of subjects: 100 subjects enrolled. Subjects must meet each of the following inclusion and exclusion criteria in order to be randomized.

Subject inclusion criteria:

* Diagnosis of PTSD, confirmed by MINI and CAPS
* Age 19 or older
* No substance abuse/dependence for the previous 4 weeks (except for nicotine and caffeine)
* Free of psychotropic medication for 2 weeks (except 4 weeks for fluoxetine)
* Clinically normal physical and laboratory examination (lab profile listed below). Liver function tests (LFTs) up to 2.5 times the normal limit will be allowed.
* Women of childbearing potential must be using medically approved methods of birth control (such as a condom, birth control pill, Depo-Provera, or diaphragm with spermicides)
* Signed informed consent
* Male or female, any race or ethnic origin

Exclusion criteria:

* Lifetime history of bipolar I, psychotic, or cognitive disorders
* Actively suicidal, homicidal, or psychotic
* History of sensitivity to mirtazapine
* Unstable general medical conditions
* Score 6 on Question #10 of MADRS regarding suicidal ideation
* Women who are pregnant, planning to become pregnant or breastfeed during the study

Exit Criteria (One needed to exit):

* Completion of the study
* Severe and intolerable side effects to mirtazapine/placebo treatment
* Acute development of suicidal ideation, homicidal ideation or psychotic symptoms
* Symptoms worsen (Score of 7 (very much worse) on CGI-I.
* Participant's explicit request to exit the study
* The need for additional psychotropic drugs, other than the study drug or adjunctive medication as specified in the protocol, for the control of the subjects psychiatric symptoms.
* The subject becomes pregnant during the course of the study.
* Investigator's judgment that it is no longer in the best interest of the patient to continue in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD, confirmed by Mini-International Neuropsychiatric Interview (MINI) and CAPS
* Age 19 or older
* No substance abuse/dependence for the previous 4 weeks (except for nicotine and caffeine)
* Free of psychotropic medication for 2 weeks (except 4 weeks for fluoxetine)
* Clinically normal physical and laboratory examination (lab profile listed below). LFTs up to 2.5 times the normal limit will be allowed.
* Women of childbearing potential must be using medically approved methods of birth control (such as a condom, birth control pill, Depo-Provera, or diaphragm with spermicides)
* Signed informed consent
* Male or female, any race or ethnic origin

Exclusion Criteria:

* Lifetime history of bipolar I, psychotic, or cognitive disorders
* Actively suicidal, homicidal, or psychotic
* History of sensitivity to mirtazapine
* Unstable general medical conditions
* Score 6 on Question #10 of MADRS regarding suicidal ideation
* Women who are pregnant, planning to become pregnant or breastfeed during the study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-04; Primary Completion 2011-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori L Davis, MD AB, Principal Investigator — Tuscaloosa VAMC
Locations (1):
- Tuscaloosa VAMC, Tuscaloosa, Alabama, United States

REFERENCES:
- [Derived] Davis LL, Pilkinton P, Lin C, Parker P, Estes S, Bartolucci A. A Randomized, Placebo-Controlled Trial of Mirtazapine for the Treatment of Posttraumatic Stress Disorder in Veterans. J Clin Psychiatry. 2020 Oct 20;81(6):20m13267. doi: 10.4088/JCP.20m13267. PMID 33084254
- See also: VA Medical Center — http://www.research.va.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Tuscaloosa and Birmingham VA Medical Centers between April 2006 and November 2010.
Pre-assignment Details: Prior to randomization, participants signed informed consent, were assessed to have met eligibility criteria including free of psychotropic medications for the previous two weeks (4 weeks for fluoxetine) prior to randomization.
Groups:
- Mirtazapine: Mirtazapine up to 45mg/qhs (three 15mg pills) as tolerated.
- Placebo: Placebo up to three pills qhs
Period: Overall Study
Arm/Group | Mirtazapine | Placebo
Started | 39 | 39
Completed | 31 | 30
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 6 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Relocation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Seventy-three (94%) were male; mean age 38.1 +/- 9.5 (SD) years in placebo group and 37.7 +/- 10.3 (SD) in mirtazapine group.
Groups:
- Mirtazapine: Mirtazapine up to 45 mg/qhs as tolerated
- Placebo: Placebo up to three tablets qhs
- Total: Total of all reporting groups
Arm/Group | Mirtazapine | Placebo | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (10.3) | 38.1 (9.5) | 37.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 37 | 36 | 73
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Structured Interview of Posttraumatic Stress Disorder (SIP)
Description: Structured Interview of Posttraumatic Stress Disorder (SIP) is a 17-item clinician-administered scale for PTSD based on Diagnostic Statistical Manual-IV criteria. The SIP has excellent test-retest reliability (0.89; p=.00001), and internal consistency (Conbach α of 0.80). The SIP showed significant correlations with the DTS (r=0.67, p=.0001) and the Impact of Event Scale (r=0.49 p=.0001). Relative to the SCID diagnosis of PTSD, sensitivity, specificity, positive predictive value, negative predictive value, and efficiency values were 100% for all indices using a score of 20 on the SIP. Items are scored on a scale from 0-4 which are summed to yield a total score ranging from 0 to 68 (higher score means more symptomatic or worse outcome). A symptom is counted as positive if it is at least a 2 (moderate).
Time Frame: Primary outcome is measured at baseline and week 8 (primary endpoint) with primary outcome change scores calculated as week 8 minus baseline score.
Population: Randomized, took at least one dose of study medication, and returned for at least one visit post-randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mirtazapine: Mirtazapine up to 45mg/qhs as tolerated
- Placebo: Placebo up to 3 tablets qhs
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 37 | 34
units on a scale | -7.61 (9.89) | -5.83 (7.41)

ADVERSE EVENTS:
Time Frame: For the duration of the 8-week study.
Description: All adverse events were collected. Adverse events were based on participant self report. Type of adverse event is not specified in final report.
Arm/Group | Mirtazapine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 22/39 | 24/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirtazapine (N=39) | Placebo (N=39)
Any Adverse Event (General disorders) | 22 (22) | 24 (24)

LIMITATIONS AND CAVEATS:
Small sample of predominantly male combat veterans limits generalizability of findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes